CLINICAL TRIAL: NCT06467149
Title: Comparison of Frailty Screening Performance and Predictive Validity of Adverse Health Outcomes in Breast Cancer Patients Using Frailty Screening Tools
Acronym: frailty
Status: Recruiting | Type: Observational
Sponsor: Ju Qiu (Other)
Collaborators: Ministry of Education, China (Other Government)
Responsible Party: Sponsor-Investigator, Ju Qiu, lecturer., Chongqing Medical University
Organization: Chongqing Medical University (Other)
Other Study IDs: qiujuchongyi; he Humanities and Social Scien (Other: Ministry of Education of China)
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Frailty Syndrome
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- To select a suitable frailty screening scale for future frailty screening of breast cancer patients: Only basic inquiries and measurements are performed on the patient, without any intervention.

SUMMARY:
This study uses the Physical Frailty Phenotype (PFP) as the diagnostic criterion for frailty and aims to explore the frailty screening scale FRAIL (The FRAIL Scale), Tilburg Frailty Index (TFI) and geriatric screening. Screening performance of Tool-8 (Geriatric-8, G-8) in breast cancer patients, to compare the predictive validity of different frailty screening scales for adverse health outcomes in breast cancer patients, and to select appropriate frailty screening methods for breast cancer patients in my country Screening scale.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of breast cancer
* Age ≥50 years old
* the treatment plan discussed by MDT includes surgery and chemotherapy
* can walk on their own (with the assistance of walking aids)

Exclusion Criteria:

* Communication disorders
* Mental disorders that can't cooperate normally
* Combined with other malignant tumours
* Terminal stage of the disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical assessment and data collection of older adults over 50 years of age with breast cancer diagnosed at a tertiary hospital in China, with no comorbidities of other malignancies.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-08-12 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Falls | From 2023.8~2025.12.
  one or more falls due to various reasons between the diagnosis of breast cancer and the second follow-up period.Does not use any scale, is a dichotomous variable with a fall score of "1" and a no fall score of "0".
Unplanned hospitalisation | 2023.8~2025.12.
  hospitalisation after doctor's diagnosis and hospitalisation for more than one day after diagnosis of breast cancer up to the second follow-up period, except for treatment nodes such as surgery and chemotherapy.No scale is used, it is a dichotomous variable with a score of "1" for unplanned hospitalisation and a score of "0" for non-occurrence.
Disability | From 2023.8~2025.12.
  Activities of daily living (ADL) were assessed using the Barthel Index (BI).The present study defined the development of disability as a decrease in scores on at least one scale entry in the BI scale from six months earlier
Depression | From 2023.8~2025.12.
  Depression screening was performed using the Geriatric Depression Scales-5 (GDS-5). The options for each entry were "yes" or "no". Entry 1 was scored 0 points for "yes" and 1 point for "no", and entries 2 to 5 were scored 1 point for "yes" and 0 points for "no". The answer "yes" for entries 2 to 5 is 1 point, and the answer "no" is 0 points. The total score ranged from 0 to 5, with a score of ≥2 indicating the presence of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Na kong, Principal Investigator — Tutor
Locations (1):
- Ju Qiu, Chongqing, China

IPD SHARING:
Plan to Share IPD: No
The study promises to keep the confidentiality of the patient, unless there is a special need, and the patient's consent should be obtained.